CLINICAL TRIAL: NCT04821700
Title: Carotid Artery Atherosclerosis in Ischemic Stroke Patients With Atrial Fibrillation.(Atrial Fibrillation and Carotid Atherosclerosis in Ischemic Stroke Patients- AFCAS)
Brief Title: Atrial Fibrillation and Carotid Atherosclerosis in Ischemic Stroke Patients-(AFCAS)
Acronym: AFCAS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, George Ntaios, Associate Professor, University of Thessaly
Other Study IDs: AFCAS 2021
Record Dates: First submitted 2021-03-21; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Ischemic Stroke; Atrial Fibrillation; Carotid Stenosis
Keywords: Ischemic Stroke; Atrial fibrillation; carotid stenosis; atherosclerosis
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation; Carotid Stenosis; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Carotid stenosis: Ischemic stroke patients with atrial fibrillation and carotid stenosis
  Interventions: Biological: Carotid Stenosis
- Patients without Carotid stenosis: Ischemic stroke patients with atrial fibrillation without carotid stenosis

INTERVENTIONS:
Biological: Carotid Stenosis — To investigate if the concurrent presence of carotid stenosis has any effect on future outcomes of patients with ischemic stroke and atrial fibrillation
  Groups: Patients with Carotid stenosis

SUMMARY:
The main aim of the study is to investigate the prevalence and characteristics of ischemic stroke patients with atrial fibrillation and concurrent carotid atherosclerosis. Additionally, this study will investigate the effect of concurrent carotid atherosclerosis on the outcomes of recurrent stroke, myocardial infarction and death during follow-up

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization due to ischemic stroke
* Atrial fibrillation
* Αny type of carotid vascular imaging

Exclusion Criteria:

* Intracerebral haemorrhage on admission
* Haemorrhagic transformation on admission

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Ischemic Stroke patients with atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-03-25 (Estimated); Study Completion 2021-04-05 (Estimated)

PRIMARY OUTCOMES:
Stroke recurrence | From date of randomization until the date of stroke recurrence, assessed up to 60 months
Myocardial infarction | From date of randomization until the date of myocardial infarction, assessed up to 60 months
Death during follow-up | From date of randomization until the date of death from any cause, assessed up to 60 months

SECONDARY OUTCOMES:
modified Rankin Scale at 3 months | 3 months
  mRS: modified Rankin Scale; 0=No symptoms at all; 1=No significant disability despite symptoms: able to carry out all usual duties and activities; 2=Slight disability: unable to carry out all previous activities, but able to look after own affairs without assistance; 3= Moderate disability: requiring some help, but able to walk without assistance; 4=Moderately severe disability: unable to walk without assistance and unable to attend to own bodily needs without assistance; 5=Severe disability: bedridden, incontinent and requiring constant nursing care and attention; 6=Dead

CONTACTS AND LOCATIONS:
Locations (1):
- Medical School, University of Thessaly, Larissa University Hospital, Larissa, Greece